CLINICAL TRIAL: NCT05128669
Title: Randomized Controlled Trial of Child and Parent-directed Individualized Psychotherapy (CPIP) for Neglected Children With Internalizing Disorders
Brief Title: Child and Parent-directed Individualized Psychotherapy (CPIP)
Acronym: AMIS-II-RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leipzig (Other)
Collaborators: Technische Universität Dresden (Other); Medical School Hamburg (Other); Technical University of Munich (Other)
Responsible Party: Principal Investigator, Lars White, Principal Investigator, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMIS-II-RCT; 01KR1802A (Other Grant/Funding Number: Federal Ministry of Education and Research Germany)
Record Dates: First submitted 2021-01-11; First posted 2021-11-22 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Child Neglect; Internalizing Disorder
Keywords: emotional/physical neglect; Internalizing disorders; 3 to 8-year old children
MeSH Terms: interventions — prostaglandin-inositol cyclic phosphate

STUDY DESIGN:
Intervention Model Description: 2 arms, randomized assignment to intervention group (CPIP + ECS) or control group (ECS only), single masked (outcomes assessor), multi-centre trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPIP+ECS (Experimental): CPIP is an innovative Child-Parent Individualized Psychotherapy, consisting of 25 sessions, designed by the PI and his clinical collaborators for children with internalizing disorders in the aftermath of childhood neglect. It is informed by Short-term Psychoanalytic Child Therapy (PaCT), elements of psychoanalytic parent work, videofeedback and Child-Parent Psychotherapy (CPP) and. CPIP supports the child-caregiver relationship and helps the child to resolve rigid conflictual internal representations/working models and improve interpretative and mentalizing techniques.
  ECS (Enhanced Caregiving Support) is described in other arm.
  Interventions: Procedure: CPIP; Procedure: ECS
- ECS only (Active Comparator): Enhanced Caregiving Support (ECS) will serve as the control condition provided by the Allgemeine Sozialdienst (ASD - Community Social Services) of the two participating cities. According to German law (§ 27 SGB VIII), caregivers are entitled to receive caregiving support (CS; "Hilfe zur Erziehung") in cases where the child's wellbeing is jeopardized. CS generally includes supportive work across all child-relevant systems (family, neighborhood, (pre-)school, peer group etc.). Appointed social workers and educators provide parenting counseling, family support, and intensive child support according to an individualized helping plan ("Hilfeplan"). In more severe cases, children are placed in (temporary) day-care centers, children's homes, foster families etc. Within the context of the trial, we will appoint an additional multi-systemic case manager to each case to enhance the quality of case coordination (enhanced CS; ECS). All children and families will receive ECS.
  Interventions: Procedure: ECS

INTERVENTIONS:
Procedure: CPIP — CPIP is an innovative Child-Parent Individualized Psychotherapy, consisting of 25 sessions, designed by the PI and his clinical collaborators for children with internalizing disorders in the aftermath of childhood neglect. It is informed by Short-term Psychoanalytic Child Therapy, elements of psychoanalytic parent work, videofeedback and Child-Parent Psychotherapy (CPP) and. CPIP supports the child-caregiver relationship and helps the child to resolve rigid conflictual internal representations/working models and improve interpretative and mentalizing techniques.
  Arms: CPIP+ECS
Procedure: ECS — Enhanced Caregiving Support (ECS) will serve as the control condition provided by the Allgemeine Sozialdienst (ASD - Community Social Services) of the two participating cities. According to German law (§ 27 SGB VIII), caregivers are entitled to receive caregiving support (CS; "Hilfe zur Erziehung") in cases where the child's wellbeing is jeopardized. CS generally includes supportive work across all child-relevant systems (family, neighborhood, (pre-)school, peer group etc.). Appointed social workers and educators provide parenting counseling, family support, and intensive child support according to an individualized helping plan ("Hilfeplan"). In more severe cases, children are placed in (temporary) day-care centers, children's homes, foster families etc. Within the context of the trial, we will appoint an additional multi-systemic case manager to each case to enhance the quality of case coordination (enhanced CS; ECS). All children and families will receive ECS.

SUMMARY:
With CPIP the investigators opt for a manualized modular psychotherapy designed especially to meet the needs of children with internalizing disorders that suffered or still suffer from emotional or physiological neglect. CPIP helps the child to resolve rigid conflictual internal representations/ working models by individually focusing on caregiver-child interaction, mentalization based interventions with children and caregivers and working with the therapeutic transference relationship with the child and the caregiver. Treatment sessions will take place at CAP.

Clinical hypotheses:

The main hypothesis of the study is that for children with internalizing disorders and experience of emotional / physical neglect, CPIP & enhanced caregiving support (intervention group) is superior in reducing internalizing symptoms compared to ECS alone (control group). Potential predictors of treatment response, as family context, gender and age, will be examined. Furthermore, the investigators will investigate possible treatment effects and mediating mechanisms, especially changes in DNA methylation profiles, HPA-dysregulation, cognitive-emotional styles, and emotional availability.

Additional elements: If the child additionally suffers from traumatic experiences of violence or sexual abuse, elements of Tf-CBT will be applied. Furthermore, elements of Interaction Guidance and ABC including video feedback will be applied in joint caregiver-child sessions. Treatment fidelity: Following the previous study, manualization, careful training and regular supervision will strive to ensure high treatment fidelity which will be systematically assessed in a random sample of two videotaped sessions per family.

DETAILED DESCRIPTION:
Setting: Typically, 25 weekly sessions of approximately 50 minutes; in the clinician's office, family home, or child protection service office (due to the limited compliance expected from some families to attend regular therapeutic sessions). When conducting treatment sessions in the home environment, principles of established and evidence-based home visitation programs, like SafeCare or Nurse-Family Partnership Program will be applied.

Therapeutic elements: Reflective developmental guidance, modeling appropriate emotional availability, understanding of the meaning and function of the symptoms within relationships together with the caregivers, identifying and labeling feelings and actions, creation of a "neglect narrative" (parallel to a trauma narrative) and conflict interpretation together with the child.

Three treatment phases: Session 1-5: Building of a working alliance, assessment of family/individual problems and resources, focus formulation; Sessions 6-20: Therapeutic work on the focus; Session 21 to 25: Detachment of the working alliance, summarizing, concluding, fostering future development.

Therapeutic strategy: The inner conflict which is currently most pressing and actively determining the child's symptoms as well as jeopardizing mental development in the present will be identified and formulated during the first 5 sessions together with the caregivers and the child (therapeutic "focus"). The following treatment phase concentrates on the jointly identified problem/conflict that has been aggregated in the focus formulation. The setting will vary (number of parent-only, child-only, and caregiver-child sessions) as a function of whether the focus predominantly lies in the interpersonal (caregiver-child interaction) or intrapersonal realm.

Control Condition: Enhanced Caregiving Support (ECS) will serve as the control condition provided by the Allgemeine Sozialdienst (ASD - Community Social Services) of the two participating cities. According to German law (§ 27 SGB VIII), caregivers are entitled to receive caregiving support (CS; "Hilfe zur Erziehung") in cases where the child's wellbeing is jeopardized. CS generally includes supportive work across all child-relevant systems (family, neighborhood, (pre-)school, peer group etc.). Appointed social workers and educators provide parenting counseling, family support, and intensive child support according to an individualized helping plan ("Hilfeplan"). In more severe cases, children are placed in (temporary) day-care centers, children's homes, foster families etc. Within the context of the trial, the investigators will appoint an additional multi-systemic case manager to each case to enhance the quality of case coordination (enhanced CS; ECS). All children and families will receive ECS. the investigators will compare children receiving CPIP plus ECS to children receiving ECS only.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for registration:

  * Age 3 to 8
  * Sufficiently stable psychosocial situation of the child for potential participation in the study
  * Written informed consent of the patient's parents or legal guardian
  * Informed oral consent of children (from 6 years)
  * Release from professional secrecy Teacher / educator
  * Positive pre-screening for internalizing symptoms
* Inclusion criteria for randomisation:

  * Confirmation that the child's psychosocial situation is sufficiently stable to participate in the study
  * physical/emotional neglect
  * DSM-5 internalizing disorder

Exclusion Criteria:

* Exclusion criteria for registration:

  * limited language skills of children or caregivers (caregiver: if communication severely impeded despite translators)
  * unresolved custody dispute
  * concurrent intensive psychotherapy of >3 months duration
  * participation of the child in other interventional trials
* Exclusion criteria for randomisation:

  * IQ < 70
  * autism or psychosis/schizophrenia spectrum disorder of the child

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2020-07-21 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-03-20 (Estimated)

PRIMARY OUTCOMES:
Assess superiority of CPIP in addition to Enhanced Caregiving Support (ECS) as compared to ECS alone. | The primary efficacy endpoint is taken 13 months after randomisation
  We assume superiority of CPIP & ECS compared to ECS alone in reducing internalizing symptoms of participating children. The Child Behavior Checklist 4-18 (CBCL 4-18) - a well-established internationally used questionnaire that reliably and validly captures child internalizing symptoms. The primary efficacy endpoint (pEP) is the CBCL 4-18 internalizing symptoms score (IntS), rated by the primary caregiver at t3 (post-treatment).
  The scale ranges from 0-62 with higher scores indicating worse outcomes.

SECONDARY OUTCOMES:
caregiver-rated internalizing symptoms for mid/long-term effects | 13 months after randomisation
  Caregiver-rated IntS using Child Behavior Checklist (CBCL 4-18) at t4 to assess mid/long-term effects. The scale ranges from 0-62 with higher scores indicating worse outcomes.
internalizing symptoms in clinical interviews | within 4 weeks before randomisation + 7 and 13 months after randomisation
  IntS for depression and anxiety assessed using the Preschool Age Psychiatric Assessment (PAPA), administered to caregivers by trained Masters-level staff
teacher-rated internalizing symptoms | within 4 weeks before randomisation + 7 and 13 months after randomisation
  (Nursery-)teacher-rated IntS using Teacher Report Form (TRF 4-18). The scale ranges from 0-70 with higher scores indicating worse outcomes.
secondary caregiver-rated internalizing symptoms | within 4 weeks before randomisation + 7 and 13 months after randomisation
  Secondary caregiver-rated IntS using Child Behavior Checklist (CBCL 4-18). The scale ranges from 0-62 with higher scores indicating worse outcomes.
child-rated internalizing symptoms | within 4 weeks before randomisation + 7 and 13 months after randomisation
  Child self-reported internalizing symptoms using Berkeley Puppet Interview. The scale ranges from 1-182 with higher scores indicating better outcomes.
Externalizing symptoms | within 4 weeks before randomisation + 7 and 13 months after randomisation
  Externalizing symptoms (ExtS) rated by caregivers and teachers using the Child Behavior Checklist (CBCL 4-18), Teacher-report Form (TRF) and Berkeley Puppet Interview, respectively.
  The CBCL ExtS scale ranges from 0-66 with higher scores indicating worse outcomes. The TRF ExtS scale ranges from 0-68 with higher scores indicating worse outcomes.
Cognitive-emotional style/mentalizing capacity | within 4 weeks before randomisation + 7 months after randomisation
  In an exploratory fashion, the investigators will test whether the child's ability to mentalize improve after the intervention and whether improvement in this ability is a mediator of the treatment effect.
  Child's ability to mentalize assessed by the Process Scales (Hill et al., 2009) and the MacArthur Narrative Coding Manual (MNCM; Robsinson et al., 2002) using the indices for narrative coherence (range: 1-12), intentionality (range: 1-12), with higher scores indicating better outcome.
Quality of the parent-child interaction (EAS) | within 4 weeks before randomisation + 7 months after randomisation
  In an exploratory fashion, the investigators will test whether the quality of parent-child interaction improve after the intervention and whether this improvement in interaction quality is a mediator of the treatment effect.
  Quality of the parent-child interaction assessed by the Emotional Availability Scales (EAS), specifically four caregiver scales (1. sensitivity, 2. structuring, 3. nonintrusiveness, and 4. nonhostility) and two child scales (1.responsiveness to mother and 2. involvement of mother). Codes on the scales range from 1 to 7, with higher scores indicating better outcome.
Cortisol secretion | within 4 weeks before randomisation + 3.5 months after randomisation + 7 and 13 months after randomisation
  hair cortisol concentrations (HCC) in the first 3 cm scalp hair segment at posterior vertex (~cumulative secretion over last 3 months)
Polygenic epigenetic risk scores | within 4 weeks before randomisation + 7 months after randomisation
  changes in DNA methylation profiles
Adherence to CPIP interventions | 7 months after randomisation
  number of sessions attended by primary caregiver and by child for secondary/sensitivity analyses
Feasibility-related endpoints - Acceptability of CPIP rated by caregivers/ parents | 7 months after randomisation
  Acceptability of CPIP rated by caregivers/ parents using Treatment evaluation questionnaire (Fragebogen zur Beurteilung der Behandlung - FBB)
Feasibility-related endpoints - Acceptability of CPIP rated by children | 7 months after randomisation
  Acceptability of CPIP rated by children: Items derived from the German version of Therapeutic Alliance Scales for Children (TASC)
Feasibility-related endpoints - Acceptability of CPIP rated by therapists | 7 months after randomisation
  Acceptability of CPIP rated by caregivers/ parents using Treatment evaluation questionnaire (Fragebogen zur Beurteilung der Behandlung - FBB)
Feasibility-related endpoints - CPIP retention rates | 7 months after randomisation
  Acceptability of CPIP - retention rates. We expect a high rate of retention until end of the intervention.
Feasibility-related endpoints - Adherence to CPIP interventions | 7 months after randomisation
  Adherence to CPIP interventions: coding of session videos using a Q-sort rating

CONTACTS AND LOCATIONS:
Overall Officials: Kai von Klitzing, Prof. Dr., Study Chair — University of Leipzig, Child and Adolescent Psychiatry
Locations (2):
- Germany (2):
  - University of Leipzig - Department of Child and Adolescent Psychiatry, Leipzig
  - Klinikum Rechts der Isar der Technischen Universität München- Lehrstuhl für Sozialpädiatrie, München

IPD SHARING:
Plan to Share IPD: Yes
After publication of the primary objective, published data might be provided to interested scientists on request (e.g. for meta-analyses, health related registers or other scientific questions) in an anonymized way within 5 years, if the members of the AMIS-II-trial group agree.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: after publication within 5 years
Access Criteria: direct inquiry to coordinating investigators